CLINICAL TRIAL: NCT02561663
Title: A Randomized, Double-blind, Placebo Controlled, Crossover Study to Determine the Effect of 5g Egg Protein Hydrolysate (NWT-03) on Arterial Stiffness, Microcirculation and Blood Pressure in Otherwise Healthy Subjects With Metabolic Syndrome
Brief Title: NWT03 and Arterial Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newtricious R&D BV (Industry)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: NWT-03 Pivotal 2
Record Dates: First submitted 2015-07-17; First posted 2015-09-28 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Metabolic Syndrome
Keywords: microcirculation; blood pressure; pulse wave analysis; pulse wave velocity
MeSH Terms: conditions — Metabolic Syndrome | interventions — NWT-03

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NWT-03, followed by placebo (Experimental): Dietary Supplement: NWT-03, an egg-white protein hydrolysate For placebo comparator, a combination of sweetener + aroma, which was equal to the combination used in the intervention period, was given Dietary Supplement: Placebo A combination of sweetener + aroma , which was equal to the combination used in the intervention period, was given.
  Interventions: Dietary Supplement: NWT-03, an egg-white protein hydrolysate; Other: Placebo
- Placebo, followed by NWT-03 (Experimental): Dietary Supplement: NWT-03, an egg-white protein hydrolysate For placebo comparator, a combination of sweetener + aroma, which was equal to the combination used in the intervention period, was given Dietary Supplement: Placebo A combination of sweetener + aroma , which was equal to the combination used in the intervention period, was given.
  Interventions: Dietary Supplement: NWT-03, an egg-white protein hydrolysate; Other: Placebo

INTERVENTIONS:
Dietary Supplement: NWT-03, an egg-white protein hydrolysate — egg-white protein hydrolysate
Other: Placebo

SUMMARY:
Rationale: Subjects with the metabolic syndrome have an increased risk of developing cardiovascular disease and a twofold risk of developing hypertension. A functional food ingredient with the ability to improve arterial stiffness, microcirculation and/or the ability to reduce blood pressure could potentially contribute to the delay or prevention of a range of cardiovascular diseases and could provide additional complimentary alternatives to pharmacological and lifestyle based interventions in the maintenance of cardiovascular health.

Objective: To assess the acute (2h) and short term (2 days and 4 week) effects of daily administration of 5g of NWT03 (an egg-protein hydrolysate) on carotid-radial Pulse Wave Velocity (cr-PWV). Secondary objectives are to assess its effects on carotid-femoral PWV, characteristics of microcirculation, systolic and diastolic blood pressure, lipid and lipoprotein metabolism, glucose metabolism and incretins.

Study design: Investigators propose to carry out a randomized, double-blind, placebo controlled crossover study.

Study population: Eligible subjects will be male or female, non-smokers between 18-75 years of age and will be otherwise healthy, but meeting at least three criteria of the Metabolic Syndrome (MetS). It is estimated that 80 otherwise healthy subjects with MetS will be randomised, to result in a minimum of 72 evaluable subjects (drop out maximal 10%) at the end of the study.

Intervention: Subjects will be randomly allocated to receive 5g of NWT-03 and placebo, once daily, on separate occasions, for a period of 4 weeks and with a washout period between the two interventions of typically 4 weeks. However, this period may be shortened by 2 weeks or extended by 8 weeks, depending on the availability of the subject. Total study duration will be 10 - 16 weeks, depending on the duration of the washout period.

Main study parameters/endpoints: Measurements will be performed at the start and end of each 4-week intervention period. Effects of NWT-03 supplementation will be calculated as the absolute differences between values obtained at each period. The main study endpoint is the change in cr-PWV.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Before the study starts, subjects will be screened to determine eligibility during a screening visit. During this visit, body weight, height, waist circumference and blood pressure will be measured and a venous blood sample (10 mL) will be collected. During the study, subjects will receive NWT-03 and placebo powders in random order and are asked to consume it on a daily basis. At visits 2, 3, 4, 5, 6 and 7 (days 0, 2, 27, 56, 58 and 83 of the study), cr-PWV, cf-PWV and office blood pressure will be recorded. A fundus photograph and a blood sample (20mL) will be taken in fasting condition. 2 hours after intake of the designated study product cr-PWV, cf-PWV and office blood pressure will again be measured and another fundus photograph will be taken. Additionally, a blood sample (20 mL) will be collected. Thus, in total 270 mL blood will be drawn. A pregnancy test will be taken in females of childbearing potential at visits 2 and 5. Subjects will be asked to fill out a food frequency questionnaire and to provide a spot urine sample at visits 4 and 7. Furthermore, subjects will be asked to keep a study diary throughout the duration of the study. Total time investment for the subjects will be approximately 19 hours. Apart from bruises or hematoma, rarely induced by blood sampling, no risks are associated with participation in this study.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrolment into the study, subjects must;

1. Be able to give written informed consent,
2. Be between 18 and 75 years of age,
3. Be in generally good health as determined by the investigator,
4. Be non-smokers
5. Have a stable body weight (< 5% change) in the 3 months prior to study entry,
6. Meet the harmonized criteria for the presence of Metabolic Syndrome as agreed by the International Diabetes Federation (IDF), National Heart Lung and Blood Institute, American Heart Association, World Heart Federation, International Atherosclerosis Society and International Association for the Study of Obesity [2], and defined as having at least three of the five following risk factors:

   * Central obesity (waist circumference >94cms in males or > 80cms in females) or having a BMI > 30 kg/m2
   * Raised triglycerides (>1.7 mmol/L (150mg/dL)
   * Reduced HDL cholesterol [<1.03mmol/L (40mg/dL) in males, <1.29mmol/L (50mg/dL) in females]
   * Raised fasting plasma glucose > 5.6mmol/L (100mg/dL)
   * Raised blood pressure (systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg)

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

1. Are less than 18 years of age or over 75 years of age,
2. Females who are pregnant, breast feeding or who may wish to become pregnant during the study,
3. Are hypersensitive to any of the components of the test product (i.e. egg protein),
4. Have a significant acute or chronic coexisting illness such as cardiovascular disease, chronic kidney disease (CKD), gastrointestinal disorder, endocrinological disorder, immunological disorder, metabolic disease or any condition which contraindicates, in the investigators judgement, entry to the study,
5. Having a condition or have taken a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include diuretics, blood pressure lowering medication and medication otherwise interfering with renin-angiotensin-aldosterone system (RAAS), such as ACE-inhibitors, angiotensin receptor blockers, direct renin inhibitors or aldosterone receptor inhibitor and cholesterol lowering agents such as statins.
6. Are taking non-steroidal anti-inflammatory drugs (NSAIDs) within 2 weeks of baseline visit or for the duration of the trial,
7. Suffer from diabetes mellitus, either type I and type II,
8. Consume more than the recommended alcohol guidelines i.e. >21 alcohol units/week for males and >14 units/week for females,
9. History of illicit drug use,
10. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial,
11. Subjects may not be receiving treatment involving experimental drugs,
12. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study or if the subject has donated blood, at a blood bank, within a period of 8 weeks prior to the start of the study.
13. Have a malignant disease or any concomitant end-stage organ disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in carotid-radial pulse wave velocity (cr-PWV) | 2 hours, 2 days and 4 weeks
  Assess the acute (2 hours) and short term (2 days and 4 week) effects of daily administration of 5g of NWT-03 on carotid radial Pulse Wave Velocity (cr-PWV)

SECONDARY OUTCOMES:
Change in carotid-femoral Pulse Wave Velocity (cf-PWV) | 2 hours, 2 days and 4 weeks
  Assess the acute (2 hours) and short term (2 days and 4 week) effects of daily administration of 5g of NWT-03 on carotid femoral Pulse Wave Velocity (cf-PWV)
Change in characteristics of microcirculation as measured by fundus photography | 2 hours, 2 days and 4 weeks
  Assess the acute (2 hours) and short term (2 days and 4 week) effects of daily administration of 5g of NWT-03 on characteristics of microcirculation as measured by fundus photography
Change in Systolic Blood Pressure | 2 hours, 2 days and 4 weeks
  Assess the acute (2 hours) and short term (2 days and 4 week) effects of daily administration of 5g of NWT-03 on Systolic Blood Pressure
Change in Diastolic Blood Pressure | 2 hours, 2 days and 4 weeks
  Assess the acute (2 hours) and short term (2 days and 4 week) effects of daily administration of 5g of NWT-03 on Diastolic Blood Pressure
Change in incretins | 4 weeks
  Assess the short term (4 weeks) effects of daily administration of 5g NWT-03 on incretins (GLP-1, GLP-2, PYY)
Change in serum HDL cholesterol concentration | 4 weeks
  Assess the short term (4 weeks) effects of daily administration of 5g NWT-03 on serum HDL cholesterol concentration
Change in serum total cholesterol concentration | 4 weeks
  Assess the short term (4 weeks) effects of daily administration of 5g NWT-03 on serum total cholesterol concentration
Change in serum LDL cholesterol concentration | 4 weeks
  Assess the short term (4 weeks) effects of daily administration of 5g NWT-03 on serum LDL cholesterol concentration
Change in serum triacylglycerol concentration | 4 weeks
  Assess the short term (4 weeks) effects of daily administration of 5g NWT-03 on serum triacylglycerol concentration
Change in glucose concentration | 4 weeks
  Assess the short term (4 weeks) effects of daily administration of 5g NWT-03 on glucose concentration
Change in insulin concentration | 4 weeks
  Assess the short term (4 weeks) effects of daily administration of 5g NWT-03 on insulin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Nijssen KMR, Joris PJ, Mensink RP, Plat J. Longer-term effects of the egg-protein hydrolysate NWT-03 on arterial stiffness and cardiometabolic risk markers in adults with metabolic syndrome: a randomized, double-blind, placebo-controlled, crossover trial. Eur J Clin Nutr. 2023 Oct;77(10):982-988. doi: 10.1038/s41430-023-01305-8. Epub 2023 Jul 7. PMID 37419971
- [Derived] Gravesteijn E, Adam JJ, Mensink RP, Winkens B, Plat J. Effects of the egg protein hydrolysate NWT-03 on cognitive function in men and women with the metabolic syndrome: a randomized, double-blind, placebo-controlled study. Nutr Neurosci. 2023 Dec;26(12):1212-1221. doi: 10.1080/1028415X.2022.2144204. Epub 2022 Nov 14. PMID 36373820